CLINICAL TRIAL: NCT03819049
Title: A Randomized, Observer-blind, First-in-Human Phase 1/2a Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Three Different Doses of VAC52416 (ExPEC10V) in Adults Aged 60 to 85 Years in Stable Health
Brief Title: A Study of Three Different Doses of VAC52416 (ExPEC10V) in Adults Aged 60 to 85 Years in Stable Health
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CR108580; VAC52416BAC1001 (Other: Janssen Research & Development, LLC); 2020-000657-27 (EudraCT Number)
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Extraintestinal Pathogenic Escherichia Coli Prevention
MeSH Terms: interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: ExPEC10V (Low Dose) (Experimental): Participants will be randomized to receive a single intramuscular (IM) injection of low dose ExPEC10V on Day 1.
  Interventions: Biological: ExPEC10V
- Cohort 1: ExPEC10V (Medium dose) (Experimental): Participants will be randomized to receive a single IM injection of medium dose ExPEC10V on Day 1.
  Interventions: Biological: ExPEC10V
- Cohort 1: ExPEC10V (High dose) (Experimental): Participants will be randomized to receive a single IM injection of high dose ExPEC10V on Day 1.
  Interventions: Biological: ExPEC10V
- Cohort 1: ExPEC4V (Experimental): Participants will be randomized to receive a single IM injection of ExPEC4V on Day 1.
  Interventions: Biological: ExPEC4V
- Cohort 1: Prevnar 13 (Experimental): Participants will be randomized to receive a single IM injection of Prevnar 13 on Day 1.
  Interventions: Biological: Prevnar 13
- Cohort 2: ExPEC10V (Experimental): Participants will be randomized to receive a single IM injection of selected dose of ExPEC10V on Day 1. The ExPEC10V dose used in Cohort 2 will be based on the primary analysis (Day 30) results of Cohort 1.
  Interventions: Biological: ExPEC10V
- Cohort 2: Placebo (Placebo Comparator): Participants will be randomized to receive a single IM injection of matching placebo on Day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ExPEC10V — Participants will receive a single IM injection of ExPEC10V (1 of 3 doses [low or medium or high]) in Cohort 1 and ExPEC10V selected dose (based on the primary analysis results of Cohort 1) in Cohort 2 on Day 1.
  Other Names: VAC52416
  Arms: Cohort 1: ExPEC10V (High dose); Cohort 1: ExPEC10V (Low Dose); Cohort 1: ExPEC10V (Medium dose); Cohort 2: ExPEC10V
Biological: ExPEC4V — Participants will receive a single IM injection of ExPEC4V on Day 1.
  Other Names: JNJ-63871860
  Arms: Cohort 1: ExPEC4V
Biological: Prevnar 13 — Participants will receive a single IM injection of Prevnar 13 on Day 1.
  Arms: Cohort 1: Prevnar 13
Biological: Placebo — Participants will receive single IM injection of matching placebo on Day 1.
  Arms: Cohort 2: Placebo

SUMMARY:
The purpose of this study is to assess the safety, reactogenicity, and immunogenicity of 3 different doses of ExPEC10V and to select the optimal dose for further clinical development (Cohort 1). Cohort 2 is aimed to expand the dataset supporting the short- and long-term safety and immunogenicity of the optimal dose of ExPEC10V, selected from the primary analysis results of Cohort 1. Cohort 2 will include participants in stable health with a history of urinary tract infection (UTI) in the past 5 years and will be included in the study to support the plan for late stage development of ExPEC vaccine.

DETAILED DESCRIPTION:
ExPEC10V (JNJ-69968054) is a 10-valent vaccine candidate in development for prevention of invasive extraintestinal pathogenic Escherichia coli (ExPEC) disease (IED) in adults 60 years of age and older. ExPEC10V consists of O-antigen polysaccharides (PSs) of the ExPEC serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B and O75 separately bioconjugate to the carrier protein, a genetically detoxified form of exotoxin A (EPA) derived from Pseudomonas aeruginosa. Since, mechanism of action of conjugate vaccines in prevention of invasive disease is not expected to be affected by antibiotic resistance mechanisms, ExPEC10V vaccine may provide protection against IED caused by drug resistant and susceptible ExPEC serotypes. The study consists of two cohorts. Cohort 1 is comprised of three periods: a screening period (28 days), an observer-blind follow-up period (181 days) with vaccination on Day 1, and an open-label long term follow up (LTFU) period (from Day 182 until 5 years [Day 1826] post-vaccination). Cohort 2 is also comprised of three periods: a screening period (28 days), a double-blind follow-up period (181 days) with vaccination on Day 1, and a double-blind LTFU period (from Day 182 until 1 years [Day 366] post-vaccination). The end of Cohort 1 is considered as the Year 5 visit (Day 1826) for the last participant. The end of Cohort 2 is considered as the Year 1 visit (Day 366) for the last participant. Key immunogenicity assessments will include the assessment of ExPEC10V and ExPEC4V serotype-specific total immunoglobulin G antibody levels elicited by the vaccine and ExPEC10V and ExPEC4V serotype-specific functional antibodies. Key safety assessments include solicited local and systemic AEs, unsolicited AEs, SAEs, physical examinations, vital sign measurements, and, for Cohort 1 only, clinical laboratory tests. The total duration of the study is up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have a body mass index (BMI) of greater than (>) 18.5 or less than 40 kilogram per meter square (kg/m^2)
* Before randomization, a woman must be: postmenopausal - A postmenopausal state is defined as no menses for 12 months without an alternative medical cause; or not intending to conceive by any methods
* Must be healthy or medically stable
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Willing and able to adhere to the lifestyle restrictions specified in this protocol
* Agrees not to donate blood until 12 weeks after receiving the study vaccine

Exclusion Criteria:

* Acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than equal to >=38.0 degree Celsius (100.4 degree Fahrenheit) within 24 hours prior to the administration of study vaccine, or, applicable for Cohort 2 only, an ongoing or suspected symptomatic urinary tract infection (UTI); enrollment at a later date is permitted (provided the screening window of 28 days is respected)
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Known allergies, hypersensitivity, or intolerance to ExPEC10V or its excipients
* Applicable for Cohort 1 only: known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the active control vaccines)
* Contraindication to intramuscular (IM) injections and blood draws example, bleeding disorders
* Abnormal function of the immune system
* Has had major psychiatric illness and/or drug substance or alcohol abuse in the past 12 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 836 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (29):
- United States (12):
  - Optimal Research, Huntsville, Alabama
  - Optimal Research, Melbourne, Florida
  - Qps-Mra, Llc, Miami, Florida
  - Optimal Research, Peoria, Illinois
  - Synexus Clinical Research US Inc, Evansville, Indiana
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Synexus Clinical Research US Inc, Richfield, Minnesota
  - Synexus Clinical Research US Inc, Manhattan, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Synexus Clinical Research US Inc, Akron, Ohio
  - Synexus Clinical Research US Inc, Columbus, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina
- Belgium (3):
  - Anima, Alken
  - ATC Pharma, Liège
  - Clinical Pharmacology Unit, Merksem
- France (6):
  - CHU Nantes, Nantes
  - Hopital Cochin, Paris
  - APHP - Hopital Bichat - Claude Bernard, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - Chu Rennes Hopital Pontchaillou, Rennes
  - CHRU Tours Hopital Bretonneau, Tours
- Netherlands (2):
  - EB Flevo Research, Almere Stad
  - PRA Health Sciences, Groningen
- Spain (6):
  - Hosp. Del Mar, Barcelona
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials\transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Fierro CA, Sarnecki M, Spiessens B, Go O, Day TA, Davies TA, van den Dobbelsteen G, Poolman J, Abbanat D, Haazen W. A randomized phase 1/2a trial of ExPEC10V vaccine in adults with a history of UTI. NPJ Vaccines. 2024 Jun 14;9(1):106. doi: 10.1038/s41541-024-00885-1. PMID 38877036

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Low Dose ExPEC10V: Participants aged greater than or equal to (>=) 60 to less than or equal to (<=) 85 years in stable health with or without a history of urinary tract infection (UTI) received a single 0.5 milliliter (mL) intramuscular (IM) injection of ExPEC10V low dose (88 micrograms polysaccharide per milliliter [mcg PS/mL]) on Day 1.
- Cohort 1: Medium Dose ExPEC10V: Participants aged >=60 to <= 85 years in stable health with or without a history of UTI received a single 0.5 mL IM injection of ExPEC10V medium dose (120 mcg PS/mL) on Day 1.
- Cohort 1: High Dose ExPEC10V: Participants aged >=60 to <= 85 years in stable health with or without a history of UTI received a single 0.5 mL IM injection of ExPEC10V high dose (176 mcg PS/mL) on Day 1.
- Cohort 1: ExPEC4V: Participants aged >=60 to <= 85 years in stable health with or without a history of UTI received a single 0.5 mL IM injection of ExPEC4V 40 mcg PS/mL on Day 1.
- Cohort 1: Prevnar 13: Participants aged >=60 to <= 85 years in stable health with or without a history of UTI received a single 0.5 mL IM injection of Prevnar 13 on Day 1.
- Cohort 2: ExPEC10V High Dose: Participants aged >=60 years in stable health with a history of UTI received a single 0.5 mL IM injection of ExPEC10V high dose (176 mcg PS/mL) on Day 1.
- Cohort 2: Placebo: Participants aged >=60 years in stable health with a history of UTI received a single 0.5 mL IM injection of placebo (matched to ExPEC10V high dose) on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13 | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Started | 104 | 102 | 104 | 53 | 54 | 280 | 139
Vaccinated | 104 | 102 | 104 | 52 | 54 | 278 | 138
Completed | 103 | 100 | 0 | 52 | 0 | 268 | 136
Not Completed | 1 | 2 | 104 | 1 | 54 | 12 | 3
Not completed — Lost to Follow-up | 1 | 2 | 9 | 0 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 18 | 0 | 10 | 9 | 1
Not completed — Ongoing | 0 | 0 | 75 | 0 | 41 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Randomized but not vaccinated | 0 | 0 | 0 | 1 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants with a vaccine administration documented.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13 | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo | Total
Number analyzed (Participants) | 104 | 102 | 104 | 52 | 54 | 278 | 138 | 832
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (5.77) | 66.4 (5.17) | 65.1 (5.15) | 64.8 (4.56) | 65.9 (5.44) | 68.7 (6.16) | 69.1 (7.21) | 67.3 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 45 | 65 | 31 | 28 | 220 | 111 | 559
  Male | 45 | 57 | 39 | 21 | 26 | 58 | 27 | 273
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 15 | 4 | 7 | 38 | 17 | 113
  Not Hispanic or Latino | 85 | 85 | 86 | 46 | 47 | 237 | 117 | 703
  Unknown or Not Reported | 2 | 2 | 3 | 2 | 0 | 3 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Asian | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 10 | 10 | 13 | 3 | 4 | 7 | 4 | 51
  White | 93 | 91 | 90 | 48 | 50 | 261 | 129 | 762
  More than one race | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  BELGIUM | 0 | 0 | 0 | 0 | 0 | 40 | 24 | 64
  FRANCE | 0 | 0 | 0 | 0 | 0 | 39 | 21 | 60
  NETHERLANDS | 0 | 0 | 0 | 0 | 0 | 40 | 11 | 51
  SPAIN | 0 | 0 | 0 | 0 | 0 | 30 | 12 | 42
  UNITED STATES | 104 | 102 | 104 | 52 | 54 | 129 | 70 | 615

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 14 Days After Vaccination on Day 1
Description: Number of participants with solicited local AEs for 14 days after vaccination on Day 1 were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. Solicited local AEs were precisely defined events that participants were specifically asked about and which were noted by participants in the diary. Solicited local (injection site) AEs included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site). All solicited AEs at the injection site (local) were considered related to the study vaccine administration.
Time Frame: Up to 14 days post vaccination on Day 1 (from Day 1 up to Day 15)
Population: Full analysis set (FAS) included all randomized participants with a vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13
Number analyzed (Participants) | 104 | 102 | 104 | 52 | 54
Participants | 46 | 54 | 60 | 15 | 40

2. Primary Outcome: Cohort 1: Number of Participants With Solicited Systemic Adverse Events (AEs) Collected for 14 Days After Vaccination on Day 1
Description: Number of participants with solicited systemic AEs 14 days after vaccination on Day 1 were reported. An AE was any untoward medical occurrence in a clinical study administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. Solicited systemic AEs included fatigue, headache, nausea, fever and myalgia, for which participants were specifically questioned and which were noted by participants in their participant diary for 14 days post-vaccination (day of vaccination and the subsequent 14 days).
Time Frame: Up to 14 days post vaccination on Day 1 (from Day 1 up to Day 15)
Population: FAS included all randomized participants with a vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13
Number analyzed (Participants) | 104 | 102 | 104 | 52 | 54
Participants | 41 | 47 | 47 | 17 | 26

3. Primary Outcome: Cohort 1: Number of Participants With Unsolicited Adverse Events (AEs) up to 29 Days After Vaccination on Day 1
Description: Number of participants with unsolicited AEs up to 29 days after vaccination on Day 1 were reported. An AE was any untoward medical occurrence in a clinical study administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: Up to 29 days post vaccination on Day 1 (from Day 1 up to Day 30)
Population: FAS included all randomized participants with a vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13
Number analyzed (Participants) | 104 | 102 | 104 | 52 | 54
Participants | 25 | 21 | 23 | 9 | 15

4. Primary Outcome: Cohort 1: Number of Participants With Serious Adverse Events (SAEs) up to Day 181
Description: Number of participants with SAEs up to Day 181 were reported. An AE was any untoward medical occurrence in a clinical study administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: Day 1 (post vaccination) up to Day 181
Population: FAS included all randomized participants with a vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13
Number analyzed (Participants) | 104 | 102 | 104 | 52 | 54
Participants | 2 | 2 | 0 | 0 | 1

5. Primary Outcome: Cohort 2: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) Collected for 14 Days After Vaccination on Day 1
Description: as for outcome 1
Time Frame: Up to 14 days post vaccination on Day 1 (from Day 1 up to Day 15)
Population: FAS included all randomized participants with a vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Number analyzed (Participants) | 278 | 138
Participants | 139 | 22

6. Primary Outcome: Cohort 2: Number of Participants With Solicited Systemic Adverse Events (AEs) Collected for 14 Days After Vaccination on Day 1
Description: as for outcome 2
Time Frame: Up to 14 days post vaccination on Day 1 (from Day 1 up to Day 15)
Population: FAS included all randomized participants with a vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Number analyzed (Participants) | 278 | 138
Participants | 139 | 53

7. Primary Outcome: Cohort 2: Number of Participants With Unsolicited Adverse Events (AEs) 29 Days After Vaccination on Day 1
Description: as for outcome 3
Time Frame: Up to 29 days post vaccination on Day 1 (from Day 1 up to Day 30)
Population: FAS included all randomized participants with a vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Number analyzed (Participants) | 278 | 138
Participants | 79 | 36

8. Primary Outcome: Cohort 2: Number of Participants With Serious Adverse Events (SAEs) up to Day 181
Description: as for outcome 4
Time Frame: Day 1 (post vaccination) up to Day 181
Population: FAS included all randomized participants with a vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Number analyzed (Participants) | 278 | 138
Participants | 9 | 6

9. Primary Outcome: Cohort 1: Geometric Mean Titers (GMTs) of Serotype-specific Total Immunoglobulin G (IgG) Serum Antibodies as Measured by Multiplex Electrochemiluminescent (ECL) Based Immunoassay on Day 15
Description: GMTs of serotype-specific total IgG serum antibodies as measured by multiplex ECL based immunoassay were reported. GMTs for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and exotoxin protein A (EPA) were determined in serum from collected blood samples.
Time Frame: Day 15
Population: Per-protocol immunogenicity (PPI) analysis set included all randomized and vaccinated participants, for whom immunogenicity data were available excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure and "n" (number analyzed) signifies those participants who were evaluable at specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13
Number analyzed (Participants) | 101 | 98 | 100 | 48 | 51
Titer
  Serotype O1A | 5350535.1 [4644976.0 to 6163266.7] | 6358232.9 [5664895.6 to 7136429.1] | 6421446.5 [5730738.4 to 7195403.5] | 6930697.9 [5823442.2 to 8248484.7] | 1606747.3 [1205014.3 to 2142411.9]
  Serotype O2 | 4873016.8 [4116237.9 to 5768931.0] | 4787891.5 [4034593.8 to 5681837.2] | 6537864.9 [5861510.6 to 7292263.1] | 6196015.3 [4955643.7 to 7746845.5] | 447845.4 [343614.9 to 583692.7]
  Serotype O4 | 2906299.6 [2339299.2 to 3610729.8] | 2778764.0 [2281609.7 to 3384246.4] | 4140729.8 [3480255.9 to 4926546.7] | 503269.8 [409184.0 to 618989.3] | 545556.7 [415552.0 to 716233.0]
  Serotype O6A | 4349111.4 [3780753.5 to 5002910.0] | 5150333.2 [4384440.1 to 6050015.8] | 5834052.6 [5130881.4 to 6633591.3] | 5051389.0 [4030377.7 to 6331051.9] | 984170.4 [805275.1 to 1202807.9]
  Serotype O8 | 5082460.4 [4435261.0 to 5824100.0] | 5605655.1 [4917150.4 to 6390564.9] | 6071895.4 [5414031.1 to 6809697.4] | 1738652.7 [1408103.9 to 2146796.9] | 1391481.0 [1093370.5 to 1770872.3]
  Serotype O15 | 5151217.3 [4393448.3 to 6039684.0] | 4635317.8 [3976055.4 to 5403891.3] | 5414798.2 [4732722.1 to 6195174.6] | 898897.3 [694569.8 to 1163333.7] | 1202517.7 [893109.0 to 1619118.0]
  Serotype O16 | 4298055.1 [3664533.7 to 5041099.1] | 3972656.6 [3378225.9 to 4671682.9] | 5675420.6 [4957603.9 to 6497170.6] | 759403.5 [619027.4 to 931612.4] | 732969.6 [586564.3 to 915917.3]
  Serotype O18A | 3532498.2 [2965791.1 to 4207492.4] | 3585987.4 [3008355.6 to 4274529.8] | 4522807.6 [3883477.9 to 5267388.9] | 1015034.0 [840693.0 to 1225529.4] | 1100583.1 [846592.3 to 1430775.0]
  Serotype O25B: number analyzed (Participants) | 101 | 98 | 99 | 48 | 51
  Serotype O25B | 1426991.8 [1113308.2 to 1829058.4] | 2265970.3 [1766736.9 to 2906273.8] | 2044257.9 [1617260.1 to 2583994.0] | 2174362.2 [1533603.8 to 3082837.4] | 267879.1 [204166.3 to 351474.3]
  Serotype O75 | 2932034.9 [2454267.7 to 3502807.9] | 3107132.4 [2627869.3 to 3673802.2] | 3963138.0 [3450884.5 to 4551430.9] | 1336846.1 [1060936.4 to 1684509.5] | 1363797.1 [1041800.4 to 1785315.7]
  Serotype EPA | 1170226.6 [829684.5 to 1650543.4] | 1496999.3 [1016330.1 to 2204999.2] | 1542536.8 [1099718.5 to 2163662.7] | 1448761.2 [868026.8 to 2418023.4] | NA [NA to 74582.5] — Geometric mean and lower limit of 95% CI could not be estimated as the value was below the lower limit of quantification (LLOQ) that is 66165.

10. Primary Outcome: Cohort 1: Geometric Mean Ratio (GMR) of Fold Changes From Baseline for Serotype Specific Antibodies as Measured by Multiplex ECL Based Immunoassay on Day 15
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by multiplex ECL based immunoassay on Day 15 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA were determined in serum from collected blood samples by multiplex ECL based immunoassay. GMR of fold change from baseline was calculated as the ratio of GMTs on Day 15 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination) and Day 15
Population: PPI analysis set included all randomized and vaccinated participants, for whom immunogenicity data were available excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure and "n" (number analyzed) signifies those participants who were evaluable at specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13
Number analyzed (Participants) | 101 | 98 | 100 | 48 | 51
Ratio
  Serotype O1A | 4.41 [3.690 to 5.259] | 5.33 [4.429 to 6.406] | 5.26 [4.381 to 6.323] | 6.00 [4.472 to 8.061] | 1.26 [1.086 to 1.452]
  Serotype O2 | 9.54 [8.014 to 11.360] | 10.05 [8.374 to 12.056] | 12.31 [10.564 to 14.334] | 12.80 [9.343 to 17.530] | 1.01 [0.953 to 1.064]
  Serotype O4 | 6.28 [5.103 to 7.718] | 5.49 [4.528 to 6.656] | 9.17 [7.610 to 11.054] | 1.06 [1.005 to 1.127] | 1.27 [1.081 to 1.491]
  Serotype O6A | 3.55 [3.039 to 4.141] | 4.48 [3.731 to 5.389] | 5.11 [4.408 to 5.918] | 4.31 [3.336 to 5.576] | 1.04 [0.990 to 1.088]
  Serotype O8 | 3.34 [2.892 to 3.855] | 3.27 [2.791 to 3.826] | 3.90 [3.362 to 4.534] | 1.07 [1.033 to 1.116] | 1.06 [0.999 to 1.128]
  Serotype O15 | 5.94 [4.966 to 7.104] | 5.32 [4.468 to 6.339] | 6.20 [5.248 to 7.329] | 1.01 [0.971 to 1.055] | 1.46 [1.223 to 1.753]
  Serotype O16 | 5.04 [4.300 to 5.912] | 4.59 [3.822 to 5.502] | 7.02 [5.904 to 8.342] | 1.11 [0.987 to 1.254] | 1.08 [1.010 to 1.155]
  Serotype O18A | 3.79 [3.220 to 4.456] | 3.64 [3.043 to 4.344] | 4.84 [4.132 to 5.675] | 1.04 [0.995 to 1.087] | 1.13 [1.027 to 1.241]
  Serotype O25B: number analyzed (Participants) | 101 | 98 | 99 | 48 | 51
  Serotype O25B | 5.80 [4.761 to 7.071] | 9.51 [7.463 to 12.126] | 8.24 [6.529 to 10.394] | 11.02 [7.889 to 15.388] | 1.02 [0.932 to 1.127]
  Serotype O75 | 2.33 [2.013 to 2.701] | 2.38 [2.055 to 2.756] | 3.06 [2.622 to 3.563] | 1.14 [1.026 to 1.274] | 1.03 [0.945 to 1.131]
  Serotype EPA | 11.31 [8.61 to 14.86] | 12.31 [9.11 to 16.62] | 11.84 [9.01 to 15.55] | 12.68 [8.28 to 19.43] | 0.99 [0.97 to 1.01]

11. Primary Outcome: Cohort 1: Percentage of Participants With a Greater Than or Equal to (>=) 2-Fold and >=4-Fold Increase From Baseline in Serotype Specific Serum Antibody Titers as Measured by Multiplex ECL Based Immunoassay on Day 15
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by multiplex ECL based immunoassay on Day 15 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Day 15 for the serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA was calculated as the ratio of titer values of serum antibody on Day 15 and pre-vaccination (on day 1) that is Day 15/Day 1.
Time Frame: Baseline (Day 1, pre-vaccination) and Day 15
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13
Number analyzed (Participants) | 101 | 98 | 100 | 48 | 51
Percentage of participants
  Serotype O1A: >= 2 Fold Increase | 78.2 [68.90 to 85.82] | 84.7 [76.01 to 91.17] | 82.0 [73.05 to 88.97] | 81.3 [67.37 to 91.05] | 9.8 [3.26 to 21.41]
  Serotype O1A: >= 4 Fold Increase | 56.4 [46.20 to 66.28] | 62. [51.88 to 71.84] | 65.0 [54.82 to 74.27] | 66.7 [51.59 to 79.60] | 5.9 [1.23 to 16.24]
  Serotype O2: >= 2 Fold Increase | 93.1 [86.24 to 97.17] | 93.9 [87.15 to 97.72] | 99.0 [94.55 to 99.97] | 89.6 [77.34 to 96.53] | 0.0 [0.00 to 6.98]
  Serotype O2: >= 4 Fold Increase | 83.2 [74.42 to 89.88] | 83.7 [74.84 to 90.37] | 92.0 [84.84 to 96.48] | 81.3 [67.37 to 91.05] | 0.0 [0.00 to 6.98]
  Serotype O4: >= 2 Fold Increase | 77.2 [67.82 to 84.98] | 81.6 [72.53 to 88.74] | 91.0 [83.60 to 95.80] | 2.1 [0.05 to 11.07] | 9.8 [3.26 to 21.41]
  Serotype O4: >= 4 Fold Increase | 64.4 [54.21 to 73.64] | 63.3 [52.93 to 72.78] | 80.0 [70.82 to 87.33] | 0.0 [0.00 to 7.40] | 3.9 [0.48 to 13.46]
  Serotype O6A: >= 2 Fold Increase | 72.3 [62.48 to 80.72] | 77.6 [68.01 to 85.36] | 86.0 [77.63 to 92.13] | 77.1 [62.69 to 87.97] | 0.0 [0.00 to 6.98]
  Serotype O6A: >= 4 Fold Increase | 42.6 [32.79 to 52.81] | 53.1 [42.71 to 63.22] | 66.0 [55.85 to 75.18] | 52.1 [37.19 to 66.71] | 0.0 [0.00 to 6.98]
  Serotype O8: >= 2 Fold Increase | 73.3 [63.54 to 81.59] | 73.5 [63.59 to 81.88] | 74.0 [64.27 to 82.26] | 0.0 [0.00 to 7.40] | 3.9 [0.48 to 13.46]
  Serotype O8: >= 4 Fold Increase | 41.6 [31.86 to 51.82] | 38.8 [29.10 to 49.15] | 51.0 [40.80 to 61.14] | 0.0 [0.00 to 7.40] | 0.0 [0.00 to 6.98]
  Serotype O15: >= 2 Fold Increase | 88.1 [80.17 to 93.71] | 82.7 [73.69 to 89.56] | 87.0 [78.80 to 92.89] | 0.0 [0.00 to 7.40] | 21.6 [11.29 to 35.32]
  Serotype O15: >= 4 Fold Increase | 61.4 [51.18 to 70.91] | 63.3 [52.93 to 72.78] | 68.0 [57.92 to 76.98] | 0.0 [0.00 to 7.40] | 9.8 [3.26 to 21.41]
  Serotype O16: >= 2 Fold Increase | 86.1 [77.84 to 92.21] | 77.6 [68.01 to 85.36] | 88.0 [79.98 to 93.64] | 2.1 [0.05 to 11.07] | 2.0 [0.05 to 10.45]
  Serotype O16: >= 4 Fold Increase | 63.4 [53.19 to 72.73] | 57.1 [46.75 to 67.10] | 73.0 [63.20 to 81.39] | 2.1 [0.05 to 11.07] | 0.0 [0.00 to 6.98]
  Serotype O18A: >= 2 Fold Increase | 72.3 [62.48 to 80.72] | 71.4 [61.42 to 80.10] | 84.0 [75.32 to 90.57] | 0.0 [0.00 to 7.40] | 3.9 [0.48 to 13.46]
  Serotype O18A: >= 4 Fold Increase | 48.5 [38.45 to 58.67] | 41.8 [31.95 to 52.23] | 61.0 [50.73 to 70.60] | 0.0 [0.00 to 7.40] | 2.0 [0.05 to 10.45]
  Serotype O25B: >= 2 Fold Increase: number analyzed (Participants) | 101 | 98 | 99 | 48 | 51
  Serotype O25B: >= 2 Fold Increase | 82.2 [73.30 to 89.08] | 87.8 [79.59 to 93.51] | 84.8 [76.24 to 91.26] | 87.5 [74.75 to 95.27] | 3.9 [0.48 to 13.46]
  Serotype O25B: >= 4 Fold Increase: number analyzed (Participants) | 101 | 98 | 99 | 48 | 51
  Serotype O25B: >= 4 Fold Increase | 58.4 [48.18 to 68.14] | 75.5 [65.79 to 83.64] | 69.7 [59.65 to 78.53] | 79.2 [65.01 to 89.53] | 2.0 [0.05 to 10.45]
  Serotype O75: >= 2 Fold Increase | 50.5 [40.36 to 60.60] | 49.0 [38.74 to 59.28] | 68.0 [57.92 to 76.98] | 6.3 [1.31 to 17.20] | 2.0 [0.05 to 10.45]
  Serotype O75: >= 4 Fold Increase | 20.8 [13.36 to 30.01] | 25.5 [17.24 to 35.31] | 33.0 [23.92 to 43.12] | 4.2 [0.51 to 14.25] | 2.0 [0.05 to 10.45]
  Serotype EPA: >= 2 Fold Increase | 87.1 [79.00 to 92.96] | 83.7 [74.84 to 90.37] | 85.0 [76.47 to 91.35] | 81.3 [67.37 to 91.05] | 0.0 [0.00 to 6.98]
  Serotype EPA: >= 4 Fold Increase | 74.3 [64.60 to 82.44] | 74.5 [64.69 to 82.76] | 77.0 [67.51 to 84.83] | 72.9 [58.15 to 84.72] | 0.0 [0.00 to 6.98]

12. Primary Outcome: Cohort 1: Geometric Mean Titers (GMT) of Serotype-specific Total Immunoglobulin G (IgG) Serum Antibodies as Measured by Multiplex Opsonophagocytic Assay (MOPA) on Day 15
Description: GMTs of serotype-specific total IgG serum antibodies as measured by MOPA were reported. GMTs for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B and O75 were determined in serum from collected blood samples.
Time Frame: Day 15
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13
Number analyzed (Participants) | 101 | 98 | 100 | 48 | 51
Titer
  Serotype O1A | 654.3 [512.4 to 835.4] | 764.2 [590.3 to 989.5] | 1129.5 [842.3 to 1514.7] | 1377.3 [851.8 to 2227.0] | 244.6 [177.9 to 336.1]
  Serotype O2: number analyzed (Participants) | 101 | 96 | 99 | 48 | 51
  Serotype O2 | 5538.4 [3884.7 to 7896.2] | 5359.8 [3689.3 to 7786.7] | 12473.2 [9082.9 to 17129.0] | 9629.4 [5960.7 to 15555.9] | 363.5 [274.0 to 482.3]
  Serotype O4 | 376.3 [278.6 to 508.2] | 322.9 [239.7 to 434.9] | 505.7 [374.6 to 682.5] | 102.9 [74.1 to 142.8] | 102.5 [79.3 to 132.5]
  Serotype O6A | 1495.9 [1133.1 to 1974.8] | 2256.5 [1725.5 to 2951.0] | 2217.2 [1690.8 to 2907.6] | 2009.8 [1344.6 to 3004.0] | 720.7 [513.8 to 1010.9]
  Serotype O8 | 1249.2 [979.3 to 1593.5] | 921.5 [702.3 to 1209.1] | 1037.6 [809.7 to 1329.6] | 712.9 [527.1 to 964.3] | 931.3 [720.7 to 1203.4]
  Serotype O15: number analyzed (Participants) | 101 | 98 | 100 | 48 | 50
  Serotype O15 | 3095.1 [2194.3 to 4365.6] | 3018.4 [2093.9 to 4351.1] | 3658.5 [2528.2 to 5294.1] | 650.2 [431.5 to 979.8] | 831.9 [542.2 to 1276.2]
  Serotype O16 | 1532.2 [1092.6 to 2148.8] | 1172.2 [822.4 to 1670.8] | 1853.8 [1353.2 to 2539.6] | 216.2 [147.0 to 317.9] | 176.9 [134.4 to 232.9]
  Serotype O18A | 274.7 [202.2 to 373.2] | 276.2 [205.0 to 372.0] | 338.2 [245.3 to 466.3] | 65.7 [44.6 to 96.9] | 62.2 [42.3 to 91.6]
  Serotype O25B | 415.5 [318.4 to 542.3] | 489.5 [373.3 to 641.9] | 403.7 [312.4 to 521.6] | 382.7 [268.7 to 545.0] | 265.4 [173.1 to 406.8]
  Serotype O75: number analyzed (Participants) | 100 | 98 | 100 | 48 | 51
  Serotype O75 | 84.0 [65.8 to 107.1] | 58.0 [46.5 to 72.3] | 91.7 [66.5 to 126.5] | NA [NA to NA] — Geometric mean, lower and upper limit of 95% CI could not be estimated as the value was below the LLOQ (37). | NA [NA to 45.3] — Geometric mean and lower limit of 95% CI could not be estimated as the value was below the LLOQ (37).

13. Primary Outcome: Cohort 1: Geometric Mean Ratio (GMR) of Fold Changes From Baseline for Serotype Specific Antibodies as Measured by MOPA on Day 15
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by MOPA on Day 15 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B and O75 were determined in serum from collected blood samples by MOPA. GMR of fold change from baseline was calculated as the ratio of GMTs on Day 15 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination), Day 15
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13
Number analyzed (Participants) | 101 | 98 | 100 | 48 | 51
Ratio
  Serotype O1A | 2.67 [2.103 to 3.389] | 4.29 [3.372 to 5.469] | 6.14 [4.546 to 8.287] | 5.34 [3.533 to 8.059] | 1.18 [0.934 to 1.484]
  Serotype O2: number analyzed (Participants) | 101 | 96 | 99 | 48 | 51
  Serotype O2 | 14.39 [10.285 to 20.126] | 17.78 [12.567 to 25.168] | 30.19 [22.504 to 40.490] | 22.96 [13.310 to 39.589] | 1.06 [0.923 to 1.228]
  Serotype O4 | 3.25 [2.489 to 4.240] | 3.47 [2.723 to 4.420] | 5.47 [4.169 to 7.178] | 0.98 [0.852 to 1.127] | 1.08 [0.917 to 1.263]
  Serotype O6A | 2.30 [1.859 to 2.858] | 3.72 [2.740 to 5.046] | 3.54 [2.782 to 4.510] | 4.30 [2.840 to 6.514] | 1.18 [1.019 to 1.368]
  Serotype O8 | 1.26 [1.078 to 1.468] | 1.22 [1.107 to 1.339] | 1.15 [0.995 to 1.324] | 0.97 [0.801 to 1.170] | 1.07 [0.891 to 1.282]
  Serotype O15: number analyzed (Participants) | 100 | 97 | 100 | 48 | 50
  Serotype O15 | 4.91 [3.498 to 6.884] | 6.29 [4.285 to 9.247] | 6.87 [4.732 to 9.980] | 0.95 [0.695 to 1.289] | 1.55 [1.076 to 2.246]
  Serotype O16 | 6.58 [4.806 to 9.018] | 5.86 [4.051 to 8.485] | 10.18 [7.527 to 13.755] | 0.94 [0.795 to 1.113] | 0.97 [0.821 to 1.157]
  Serotype O18A | 4.05 [3.148 to 5.204] | 4.27 [3.192 to 5.721] | 6.20 [4.645 to 8.279] | 1.03 [0.869 to 1.217] | 1.17 [0.941 to 1.458]
  Serotype O25B | 2.34 [1.883 to 2.903] | 2.77 [2.155 to 3.557] | 2.51 [2.033 to 3.096] | 2.48 [1.830 to 3.367] | 1.44 [1.040 to 1.997]
  Serotype O75: number analyzed (Participants) | 100 | 98 | 100 | 48 | 51
  Serotype O75 | 1.92 [1.600 to 2.299] | 1.69 [1.440 to 1.991] | 2.58 [1.981 to 3.355] | 0.97 [0.879 to 1.064] | 1.03 [0.930 to 1.133]

14. Primary Outcome: Cohort 1: Percentage of Participants With a >= 2-Fold and >=4-Fold Increase in Serotype-specific Serum Antibody Titers Measured by MOPA on Day 15
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by MOPA on Day 15 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Day 15 for the serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, and O75 was calculated as the ratio of titer values of serum antibody on Day 15 and pre-vaccination (on day 1) that is, Day 15/Day 1.
Time Frame: Baseline (Day 1, pre-vaccination) and Day 15
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13
Number analyzed (Participants) | 101 | 98 | 100 | 48 | 51
Percentage of participants
  Serotype O1A: >= 2 Fold Increase | 49.5 [39.40 to 59.64] | 70.4 [60.34 to 79.21] | 72.0 [62.13 to 80.52] | 75.0 [60.40 to 86.36] | 13.7 [5.70 to 26.26]
  Serotype O1A: >= 4 Fold Increase | 28.7 [20.15 to 38.57] | 46.9 [36.78 to 57.29] | 53.0 [42.76 to 63.06] | 52.1 [37.19 to 66.71] | 3.9 [0.48 to 13.46]
  Serotype O2: >= 2 Fold Increase: number analyzed (Participants) | 101 | 96 | 99 | 48 | 51
  Serotype O2: >= 2 Fold Increase | 90.1 [82.54 to 95.15] | 86.5 [77.96 to 92.59] | 98.0 [92.89 to 99.75] | 87.5 [74.75 to 95.27] | 11.8 [4.44 to 23.87]
  Serotype O2: >= 4 Fold Increase: number analyzed (Participants) | 101 | 96 | 99 | 48 | 51
  Serotype O2: >= 4 Fold Increase | 74.3 [64.60 to 82.44] | 78.1 [68.53 to 85.92] | 88.9 [80.99 to 94.32] | 77.1 [62.69 to 87.97] | 0.0 [0.00 to 6.98]
  Serotype O4: >= 2 Fold Increase | 56.4 [46.20 to 66.28] | 60.2 [49.82 to 69.96] | 73.0 [63.20 to 81.39] | 4.2 [0.51 to 14.25] | 11.8 [4.44 to 23.87]
  Serotype O4: >= 4 Fold Increase | 33.7 [24.56 to 43.75] | 38.8 [29.10 to 49.15] | 56.0 [45.72 to 65.92] | 2.1 [0.05 to 11.07] | 3.9 [0.48 to 13.46]
  Serotype O6A: >= 2 Fold Increase | 47.5 [37.49 to 57.70] | 54.1 [43.71 to 64.20] | 63.0 [52.76 to 72.44] | 66.7 [51.59 to 79.60] | 9.8 [3.26 to 21.41]
  Serotype O6A: >= 4 Fold Increase | 23.8 [15.86 to 33.26] | 41.8 [31.95 to 52.23] | 40.0 [30.33 to 50.28] | 39.6 [25.77 to 54.73] | 2.0 [0.05 to 10.45]
  Serotype O8: >= 2 Fold Increase | 19.8 [12.54 to 28.91] | 14.3 [8.04 to 22.81] | 10.0 [4.90 to 17.62] | 6.3 [1.31 to 17.20] | 11.8 [4.44 to 23.87]
  Serotype O8: >= 4 Fold Increase | 5.9 [2.21 to 12.48] | 3.1 [0.64 to 8.69] | 4.0 [1.10 to 9.9] | 2.1 [0.05 to 11.07] | 3.9 [0.48 to 13.46]
  Serotype O15: >= 2 Fold Increase: number analyzed (Participants) | 100 | 97 | 100 | 48 | 50
  Serotype O15: >= 2 Fold Increase | 61.0 [50.73 to 70.60] | 67.0 [56.73 to 76.22] | 70.0 [60.02 to 78.76] | 12.5 [4.73 to 25.25] | 28.0 [16.23 to 42.49]
  Serotype O15: >= 4 Fold Increase: number analyzed (Participants) | 100 | 97 | 100 | 48 | 50
  Serotype O15: >= 4 Fold Increase | 41.0 [31.26 to 51.29] | 53.6 [43.19 to 63.80] | 57.0 [46.71 to 66.86] | 8.3 [2.32 to 19.9] | 14.0 [5.82 to 26.74]
  Serotype O16: >= 2 Fold Increase | 76.2 [66.74 to 84.14] | 70.4 [60.34 to 79.21] | 85.0 [76.47 to 91.35] | 8.3 [2.32 to 19.9] | 9.8 [3.26 to 21.41]
  Serotype O16: >= 4 Fold Increase | 55.4 [45.22 to 65.34] | 51.0 [40.72 to 61.26] | 76.0 [66.43 to 83.98] | 2.1 [0.05 to 11.07] | 3.9 [0.48 to 13.46]
  Serotype O18A: >= 2 Fold Increase | 69.3 [59.34 to 78.10] | 66.3 [56.07 to 75.56] | 77.0 [67.51 to 84.83] | 6.3 [1.31 to 17.20] | 7.8 [2.18 to 18.88]
  Serotype O18A: >= 4 Fold Increase | 45.5 [35.60 to 55.76] | 44.9 [34.83 to 55.28] | 58.0 [47.71 to 67.80] | 4.2 [0.51 to 14.25] | 5.9 [1.23 to 16.24]
  Serotype O25B: >= 2 Fold Increase | 47.5 [37.49 to 57.70] | 50.0 [39.73 to 60.27] | 50.0 [39.83 to 60.17] | 50.0 [35.23 to 64.77] | 15.7 [7.02 to 28.59]
  Serotype O25B: >= 4 Fold Increase | 24.8 [16.70 to 34.33] | 33.7 [24.44 to 43.93] | 31.0 [22.13 to 41.03] | 35.4 [22.16 to 50.54] | 5.9 [1.23 to 16.24]
  Serotype O75: >= 2 Fold Increase | 36.0 [26.64 to 46.21] | 28.6 [19.9 to 38.58] | 38.0 [28.48 to 48.25] | 0.0 [0.00 to 7.40] | 3.9 [0.48 to 13.46]
  Serotype O75: >= 4 Fold Increase | 16.0 [9.43 to 24.68] | 17.3 [10.44 to 26.31] | 25.0 [16.88 to 34.66] | 0.0 [0.00 to 7.40] | 0.0 [0.00 to 6.98]

15. Primary Outcome: Cohort 2: Geometric Mean Titers (GMTs) of Serotype-specific Total Immunoglobulin G (IgG) Serum Antibodies as Measured by Multiplex ECL Based Immunoassay on Day 30
Description: GMTs of serotype-specific total IgG serum antibodies as measured by multiplex ECL based immunoassay were reported. GMTs for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA were determined in serum from collected blood samples.
Time Frame: At Day 30
Population: PPI analysis set included all randomized and vaccinated participants, for whom immunogenicity data were available excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Number analyzed (Participants) | 258 | 129
Titer
  Serotype O1A | 6341302.4 [5889782.4 to 6827436.7] | 1762724.3 [1505477.9 to 2063927.4]
  Serotype O2 | 5957433.5 [5487954.2 to 6467075.6] | 749984.6 [628913.9 to 894362.5]
  Serotype O4 | 3537556.6 [3153145.2 to 3968833.1] | 805295.5 [689894.4 to 940000.1]
  Serotype O6A | 5461039.4 [4992165.2 to 5973951.2] | 1944280.6 [1664293.0 to 2271371.1]
  Serotype O8 | 6240213.6 [5782238.7 to 6734461.7] | 2315932.9 [2011986.2 to 2665796.4]
  Serotype O15 | 5724175.1 [5301709.2 to 6180305.1] | 1207724.5 [1028556.8 to 1418101.9]
  Serotype O16 | 5158063.5 [4735530.7 to 5618297.2] | 1127584.4 [1001022.6 to 1270147.7]
  Serotype O18 | 4046778.4 [3656809.6 to 4478334.1] | 1365154.9 [1196273.0 to 1557878.4]
  Serotype O25B | 2117662.8 [1843164.1 to 2433042.1] | 375570.5 [316412.1 to 445789.5]
  Serotype O75 | 3758021.3 [3419541.0 to 4130005.8] | 1577900.4 [1365705.2 to 1823065.1]
  Serotype EPA | 780539.6 [622435.7 to 978803.3] | 75018.0 [NA to 91880.8] — Lower limit of 95% CI could not be estimated as the value was below the LLOQ (66165).

16. Primary Outcome: Cohort 2: Geometric Mean Ratio (GMR) of Serotype-specific Antibodies Measured by Multiplex ECL Based Immunoassay on Day 30
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by multiplex ECL based immunoassay on Day 30 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA were determined in serum from collected blood samples by multiplex ECL based immunoassay. GMR of fold change from baseline was calculated as the ratio of GMTs on Day 30 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination) and Day 30
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Number analyzed (Participants) | 258 | 129
Ratio
  Serotype O1A | 4.40 [3.958 to 4.893] | 1.02 [0.955 to 1.095]
  Serotype O2 | 8.18 [7.255 to 9.227] | 0.98 [0.909 to 1.055]
  Serotype O4 | 5.31 [4.726 to 5.955] | 1.09 [1.014 to 1.168]
  Serotype O6A | 3.64 [3.289 to 4.019] | 1.06 [0.993 to 1.138]
  Serotype O8 | 2.92 [2.655 to 3.221] | 1.01 [0.965 to 1.058]
  Serotype O15 | 5.00 [4.483 to 5.565] | 1.02 [0.961 to 1.077]
  Serotype O16 | 5.04 [4.571 to 5.561] | 1.06 [0.993 to 1.126]
  Serotype O18 | 3.40 [3.088 to 3.754] | 1.07 [1.017 to 1.132]
  Serotype O25B | 5.59 [4.866 to 6.428] | 1.04 [0.963 to 1.115]
  Serotype O75 | 2.33 [2.136 to 2.531] | 1.04 [0.979 to 1.110]
  Serotype EPA | 8.06 [6.73 to 9.64] | 1.02 [0.97 to 1.08]

17. Primary Outcome: Cohort 2: Percentage of Participants With a >=2-Fold and >=4-Fold Increase From Baseline in Serotype Specific Serum Antibody Titers as Measured by Multiplex ECL Based Immunoassay on Day 30
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by multiplex ECL based immunoassay on Day 30 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Day 30 for the serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA was calculated as the ratio of titer values of serum antibody on Day 30 and pre-vaccination (on day 1) that is, Day 30/Day 1.
Time Frame: Baseline (Day 1, pre-vaccination) and Day 30
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Number analyzed (Participants) | 258 | 129
Percentage of participants
  Serotype O1A: >= 2 Fold Increase | 78.3 [72.76 to 83.17] | 1.6 [0.19 to 5.49]
  Serotype O1A: >= 4 Fold Increase | 54.7 [48.36 to 60.84] | 0.8 [0.02 to 4.24]
  Serotype O2: >= 2 Fold Increase | 89.1 [84.70 to 92.67] | 1.6 [0.19 to 5.49]
  Serotype O2: >= 4 Fold Increase | 77.5 [71.93 to 82.46] | 1.6 [0.19 to 5.49]
  Serotype O4: >= 2 Fold Increase | 81.4 [76.10 to 85.95] | 2.3 [0.48 to 6.65]
  Serotype O4: >= 4 Fold Increase | 58.9 [52.64 to 64.98] | 1.6 [0.19 to 5.49]
  Serotype O6A: >= 2 Fold Increase | 73.3 [67.41 to 78.56] | 2.3 [0.48 to 6.65]
  Serotype O6A: >= 4 Fold Increase | 44.2 [38.03 to 50.48] | 0.8 [0.02 to 4.24]
  Serotype O8: >= 2 Fold Increase | 64. [57.77 to 69.82] | 1.6 [0.19 to 5.49]
  Serotype O8: >= 4 Fold Increase | 38.4 [32.41 to 44.61] | 1.6 [0.19 to 5.49]
  Serotype O15: >= 2 Fold Increase | 84.1 [79.07 to 88.35] | 1.6 [0.19 to 5.49]
  Serotype O15: >= 4 Fold Increase | 58.5 [52.25 to 64.60] | 0.8 [0.02 to 4.24]
  Serotype O16: >= 2 Fold Increase | 86.0 [81.21 to 90.03] | 1.6 [0.19 to 5.49]
  Serotype O16: >= 4 Fold Increase | 62.4 [56.18 to 68.33] | 1.6 [0.19 to 5.49]
  Serotype O18: >= 2 Fold Increase | 69.0 [62.96 to 74.58] | 1.6 [0.19 to 5.49]
  Serotype O18: >= 4 Fold Increase | 43.0 [36.90 to 49.31] | 0.8 [0.02 to 4.24]
  Serotype O25B: >= 2 Fold Increase | 78.3 [72.76 to 83.17] | 2.3 [0.48 to 6.65]
  Serotype O25B: >= 4 Fold Increase | 56.6 [50.30 to 62.72] | 1.6 [0.19 to 5.49]
  Serotype O75: >= 2 Fold Increase | 51.2 [44.89 to 57.41] | 2.3 [0.48 to 6.65]
  Serotype O75: >= 4 Fold Increase | 23.6 [18.59 to 29.31] | 2.3 [0.48 to 6.65]
  Serotype EPA: >= 2 Fold Increase | 77.9 [72.34 to 82.82] | 1.6 [0.19 to 5.49]
  Serotype EPA: >= 4 Fold Increase | 65.5 [59.36 to 71.29] | 1.6 [0.19 to 5.49]

18. Primary Outcome: Cohort 2: Geometric Mean Titer (GMT) of Serotype-specific Total Immunoglobulin G (IgG) Serum Antibodies as Measured by Multiplex Opsonophagocytic Assay (MOPA) on Day 30
Description: GMTs of serotype-specific total IgG serum antibodies as measured by MOPA were reported. GMTs for each antigen serotypes O1A, O2, O4, O6A, O15, O16, O18A, O25B, and O75 were determined in serum from collected blood samples. For serotype O8 functional IgG serum antibodies were not evaluated as the assay was not able to detect vaccine-induced functional antibodies against the O8 serotype.
Time Frame: At Day 30
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Number analyzed (Participants) | 258 | 70
Titer
  Serotype O1A | 703.0 [611.1 to 808.7] | 492.4 [382.9 to 633.2]
  Serotype O2 | 3523.2 [2950.7 to 4206.7] | 502.4 [403.6 to 625.4]
  Serotype O4 | 803.9 [683.3 to 945.7] | 178.7 [138.7 to 230.4]
  Serotype O6A | 1392.6 [1196.9 to 1620.3] | 557.0 [416.8 to 744.3]
  Serotype O15 | 2773.8 [2347.4 to 3277.6] | 458.0 [338.4 to 619.9]
  Serotype O16 | 1347.0 [1132.2 to 1602.5] | 116.0 [88.0 to 152.8]
  Serotype O18 | 516.3 [446.2 to 597.3] | 168.2 [128.8 to 219.6]
  Serotype O25B | 159.8 [135.4 to 188.5] | NA [NA to 69.6] — Geometric mean and lower limit of 95% CI could not be estimated as the value was below the LLOQ (58).
  Serotype O75: number analyzed (Participants) | 257 | 69
  Serotype O75 | 201.0 [169.5 to 238.3] | 52.2 [39.2 to 69.6]

19. Primary Outcome: Cohort 2: Geometric Mean Ratio (GMR) of Fold Changes From Baseline for Serotype Specific Antibodies as Measured by MOPA on Day 30
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by MOPA on Day 30 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O15, O16, O18A, O25B and O75 were determined in serum from collected blood samples by MOPA. GMR of fold change from baseline was calculated as the ratio of GMTs on Day 30 and pre-vaccination (on Day 1). For serotype O8 functional IgG serum antibodies were not evaluated as the assay was not able to detect vaccine-induced functional antibodies against the O8 serotype.
Time Frame: Baseline (Day 1, pre-vaccination) and Day 30
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Number analyzed (Participants) | 258 | 70
Ratio
  Serotype O1A | 1.81 [1.602 to 2.054] | 1.23 [1.036 to 1.451]
  Serotype O2 | 8.04 [6.684 to 9.681] | 1.07 [0.901 to 1.265]
  Serotype O4 | 4.26 [3.607 to 5.033] | 0.98 [0.827 to 1.162]
  Serotype O6A | 2.57 [2.251 to 2.939] | 1.02 [0.870 to 1.192]
  Serotype O15 | 6.70 [5.641 to 7.958] | 1.05 [0.807 to 1.376]
  Serotype O16 | 9.68 [8.055 to 11.639] | 1.02 [0.841 to 1.227]
  Serotype O18 | 2.88 [2.482 to 3.332] | 0.93 [0.805 to 1.083]
  Serotype O25B | 2.05 [1.813 to 2.308] | 0.94 [0.841 to 1.045]
  Serotype O75: number analyzed (Participants) | 255 | 68
  Serotype O75 | 3.21 [2.744 to 3.745] | 1.18 [0.973 to 1.438]

20. Primary Outcome: Cohort 2: Percentage of Participants With a >= 2-Fold and >=4-Fold Increase in Serotype-specific Serum Antibodies Titers Measured by MOPA on Day 30
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibodies titers as measured by MOPA on Day 30 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Day 30 for the serotypes O1A, O2, O4, O6A, O15, O16, O18A, O25B and O75 was calculated as the ratio of titer values of serum antibodies on Day 30 and pre-vaccination (on day 1) that is, Day 30/Day 1. For serotype O8 functional IgG serum antibodies were not evaluated as the assay was not able to detect vaccine-induced functional antibodies against the O8 serotype.
Time Frame: Baseline (Day 1, pre-vaccination) and Day 30
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
Number analyzed (Participants) | 258 | 70
Percentage of participants
  Serotype O1A: >= 2 Fold Increase | 41.5 [35.40 to 47.75] | 22.9 [13.67 to 34.45]
  Serotype O1A: >= 4 Fold Increase | 17.8 [13.36 to 23.06] | 2.9 [0.35 to 9.94]
  Serotype O2: >= 2 Fold Increase | 81.0 [75.68 to 85.61] | 18.6 [10.28 to 29.66]
  Serotype O2: >= 4 Fold Increase | 63.6 [57.37 to 69.45] | 4.3 [0.89 to 12.02]
  Serotype O4: >= 2 Fold Increase | 64.7 [58.56 to 70.55] | 14.3 [7.07 to 24.71]
  Serotype O4: >= 4 Fold Increase | 45.7 [39.54 to 52.03] | 4.3 [0.89 to 12.02]
  Serotype O6A: >= 2 Fold Increase | 54.3 [47.97 to 60.46] | 17.1 [9.18 to 28.03]
  Serotype O6A: >= 4 Fold Increase | 32.9 [27.24 to 39.05] | 1.4 [0.04 to 7.70]
  Serotype O15: >= 2 Fold Increase | 81.4 [76.10 to 85.95] | 22.9 [13.67 to 34.45]
  Serotype O15: >= 4 Fold Increase | 62.8 [56.58 to 68.71] | 8.6 [3.21 to 17.73]
  Serotype O16: >= 2 Fold Increase | 86.0 [81.21 to 90.03] | 18.6 [10.28 to 29.66]
  Serotype O16: >= 4 Fold Increase | 70.9 [64.98 to 76.40] | 4.3 [0.89 to 12.02]
  Serotype O18: >= 2 Fold Increase | 55.8 [49.52 to 61.97] | 14.3 [7.07 to 24.71]
  Serotype O18: >= 4 Fold Increase | 34.5 [28.71 to 40.64] | 0.0 [0.00 to 5.13]
  Serotype O25B: >= 2 Fold Increase | 41.1 [35.02 to 47.36] | 5.7 [1.58 to 13.99]
  Serotype O25B: >= 4 Fold Increase | 21.3 [16.48 to 26.83] | 0.0 [0.00 to 5.13]
  Serotype O75: >= 2 Fold Increase: number analyzed (Participants) | 255 | 68
  Serotype O75: >= 2 Fold Increase | 58.4 [52.12 to 64.55] | 23.5 [14.09 to 35.38]
  Serotype O75: >= 4 Fold Increase: number analyzed (Participants) | 255 | 68
  Serotype O75: >= 4 Fold Increase | 36.9 [30.93 to 43.11] | 10.3 [4.24 to 20.07]

21. Secondary Outcome: Cohort 1: Correlation Between the Multiplex ECL-Based Immunoassay and the MOPA Functional Titers by Serotypes on Day 15
Description: Correlation between the multiplex ECL-based immunoassay and the MOPA functional titers by serotypes on Day 15 will be analyzed.
Time Frame: Day 15
Reporting Status: Not Posted, anticipated posting 2025-12

22. Secondary Outcome: Cohort 1: Geometric Mean Titers (GMTs) of Serotype-specific Total Immunoglobulin G (IgG) Serum Antibodies as Measured by Multiplex ECL Based Immunoassay on Days 30 and 181
Description: GMTs of serotype-specific total IgG serum antibodies as measured by ECL based immunoassay were reported. GMTs for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA were determined in serum from collected blood samples.
Time Frame: Days 30 and 181
Reporting Status: Not Posted, anticipated posting 2025-12

23. Secondary Outcome: Cohort 1: Percentage of Participants With a Greater Than or Equal to (>=) 2-Fold and >=4-Fold Increase From Baseline in Serotype Specific Serum Antibody Titers as Measured by Multiplex ECL Based Immunoassay on Days 30 and 181
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by multiplex ECL based immunoassay on Days 30 and 181 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Days 30 and 181 for the serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA was calculated as the ratio of titer values of serum antibody on Day 30 and Day 181 and pre-vaccination (on Day 1) that is, Day 30/Day 1 and Day 181/Day 1.
Time Frame: Day 1 (pre-vaccination) and Days 30 and 181
Reporting Status: Not Posted, anticipated posting 2025-12

24. Secondary Outcome: Cohort 1: Geometric Mean Ratio (GMR) of Serotype-specific Antibodies Measured by Multiplex ECL Based Immunoassay on Days 30 and 181
Description: GMR of fold changes from baseline for serotype specific antibodies measured by multiplex ECL based immunoassay on Days 30 and 181 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA were determined in serum from collected blood samples by ECL based immunoassay. GMR of fold change from baseline was calculated as the ratio of GMTs on Days 30 and 181 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination) and Days 30 and 181
Reporting Status: Not Posted, anticipated posting 2025-12

25. Secondary Outcome: Cohort 1: Geometric Mean Titer (GMT) of Serotype-specific Total Immunoglobulin G (IgG) Serum Antibodies as Measured by Multiplex Opsonophagocytic Assay (MOPA) on Days 30 and 181
Description: as for outcome 12
Time Frame: At Days 30 and 181
Reporting Status: Not Posted, anticipated posting 2025-12

26. Secondary Outcome: Cohort 1: Geometric Mean Ratio (GMR) of Fold Changes From Baseline for Serotype Specific Antibodies as Measured by MOPA on Days 30 and 181
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by MOPA on Days 30 and 181 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B and O75 were determined in serum from collected blood samples by MOPA. GMR of fold change from baseline was calculated as the ratio of GMTs on Days 30 and 181 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination), and Days 30 and 181
Reporting Status: Not Posted, anticipated posting 2025-12

27. Secondary Outcome: Cohort 1: Percentage of Participants With a >= 2-Fold and >=4-Fold Increase in Serotype-specific Serum Antibody Titers Measured by MOPA on Days 30 and 181
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by MOPA on Days 30 and 181 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Days 30 and 181 for the serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, and O75 was calculated as the ratio of titer values of serum antibody on Days 30 and 181 and pre-vaccination (on day 1) that is, Day 30/Day 1 and 181/Day 1.
Time Frame: Baseline (Day 1, pre-vaccination) and Days 30 and 181
Reporting Status: Not Posted, anticipated posting 2025-12

28. Secondary Outcome: Cohort 1: Number of Participants With Serious Adverse Events (SAEs) Related to Study Vaccine or Study Procedure From Day 182 up to End of Study (Day 1826)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: From Day 182 up to end of study (Day 1826)
Reporting Status: Not Posted, anticipated posting 2025-12

29. Secondary Outcome: Cohort 1: Geometric Mean Titers (GMTs) of Serotype-specific Total Immunoglobulin G (IgG) Serum Antibodies as Measured by Multiplex ECL Based Immunoassay on Days 366, 731, 1096, 1461 and 1826
Description: as for outcome 22
Time Frame: Days 366, 731, 1096, 1461 and 1826
Reporting Status: Not Posted, anticipated posting 2025-12

30. Secondary Outcome: Cohort 1: Percentage of Participants With a >=2-Fold and >=4-Fold Increase From Baseline in Serotype Specific Serum Antibody Titers as Measured by Multiplex ECL Based Immunoassay on Days 366, 731, 1096, 1461 and 1826
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by multiplex ECL based immunoassay on Days 366, 731, 1096, 1461 and 1826 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Days 366, 731, 1096, 1461 and 1826 for the serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA was calculated as the ratio of titer values of serum antibody on Days 366, 731, 1096, 1461 and 1826 and pre-vaccination (on day 1) that is, Day 366/Day 1, 731/Day 1, 1096/Day 1, 1461/Day 1 and 1826 /Day 1.
Time Frame: Baseline (Day 1, pre-vaccination) and Days 366, 731, 1096, 1461, 1826
Reporting Status: Not Posted, anticipated posting 2025-12

31. Secondary Outcome: Cohort 1: Geometric Mean Ratio (GMR) of Serotype-specific Antibodies Measured by Multiplex ECL Based Immunoassay on Days 366, 731, 1096, 1461 and 1826
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by multiplex ECL based immunoassay on Days 366, 731, 1096, 1461 and 1826 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA were determined in serum from collected blood samples by ECL based immunoassay. GMR of fold change from baseline was calculated as the ratio of GMTs on Days 366, 731, 1096, 1461 and 1826 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination) and Days 366, 731, 1096, 1461, 1826
Reporting Status: Not Posted, anticipated posting 2025-12

32. Secondary Outcome: Cohort 1: Geometric Mean Titer (GMT) of Serotype-specific Total Immunoglobulin G (IgG) Serum Antibodies as Measured by MOPA on Days 366, 731, 1096, 1461 and 1826
Description: as for outcome 12
Time Frame: Days 366, 731, 1096, 1461 and 1826
Reporting Status: Not Posted, anticipated posting 2025-12

33. Secondary Outcome: Cohort 1: Geometric Mean Ratio (GMR) of Fold Changes From Baseline for Serotype Specific Antibodies as Measured by MOPA on Days 366, 731, 1096, 1461 and 1826
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by MOPA on Days 366, 731, 1096, 1461 and 1826 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B and O75 were determined in serum from collected blood samples by MOPA. GMR of fold change from baseline was calculated as the ratio of GMTs on Days 366, 731, 1096, 1461 and 1826 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination) and Days 366, 731, 1096, 1461, 1826
Reporting Status: Not Posted, anticipated posting 2025-12

34. Secondary Outcome: Cohort 1: Percentage of Participants With a >= 2-Fold and >=4-Fold Increase in Serotype-specific Serum Antibody Titers Measured by MOPA on Days 366, 731, 1096, 1461 and 1826
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by MOPA on Days 366, 731, 1096, 1461 and 1826 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Days 366, 731, 1096, 1461 and 1826 for the serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, and O75 was calculated as the ratio of titer values of serum antibody on Days 366, 731, 1096, 1461 and 1826 and pre-vaccination (on day 1) that is, Day 366/Day 1, 731/Day 1, 1096/Day 1, 1461/Day 1 and 1826/Day 1.
Time Frame: Baseline (Day 1, pre-vaccination) and Days 366, 731, 1096, 1461, 1826
Reporting Status: Not Posted, anticipated posting 2025-12

35. Secondary Outcome: Cohort 2: Correlation Between the Multiplex ECL-Based Immunoassay and the MOPA Functional Titers by Serotype on Day 30
Description: Correlation between the multiplex ECL-based immunoassay and the MOPA functional titers by serotype on Day 30 will be analyzed.
Time Frame: At Day 30
Reporting Status: Not Posted, anticipated posting 2025-12

36. Secondary Outcome: Cohort 2: Geometric Mean Titers (GMTs) of Serotype-specific Total Immunoglobulin G (IgG) Serum Antibodies as Measured by Multiplex ECL Based Immunoassay on Days 15 and 181
Description: as for outcome 22
Time Frame: At Days 15 and 181
Reporting Status: Not Posted, anticipated posting 2025-12

37. Secondary Outcome: Cohort 2: Geometric Mean Ratio (GMR) of Serotype-specific Antibodies Measured by Multiplex ECL Based Immunoassay on Days 15 and 181
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by multiplex ECL based immunoassay on Days 15 and 181 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA were determined in serum from collected blood samples by ECL based immunoassay. GMR of fold change from baseline was calculated as the ratio of GMTs on Days 15 and 181 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination), Days 15 and 181
Reporting Status: Not Posted, anticipated posting 2025-12

38. Secondary Outcome: Cohort 2: Percentage of Participants With a >= 2-Fold and >=4-Fold Increase in Serotype-specific Serum Antibody Titers Measured by Multiplex ECL Based Immunoassay on Days 15 and 181
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by multiplex ECL based immunoassay on Days 15 and 181 were reported. The fold (>=2-fold and >=4-fold) increase from baseline to Days 15 and 181 for the serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA was calculated as the ratio of titer values of serum antibody on Days 15 and 181 and pre-vaccination (on day 1) that is Day 15/Day 1 and Day 181/Day 1.
Time Frame: Baseline (Day 1, pre-vaccination) and Days 15 and 181
Reporting Status: Not Posted, anticipated posting 2025-12

39. Secondary Outcome: Cohort 2: Geometric Mean Titers (GMTs) of Serotype-specific Antibodies Against Specified Antigens Measured by MOPA on Day 181
Description: GMTs of serotype-specific total IgG serum antibodies as measured by MOPA were reported. GMTs for each antigen serotypes O1A, O2, O4, O6A, O15, O16, O18A, O25B, and O75 were determined in serum from collected blood samples.
Time Frame: At Day 181
Reporting Status: Not Posted, anticipated posting 2025-12

40. Secondary Outcome: Cohort 2: Percentage of Participants With a >= 2-Fold and >=4-Fold Increase in Serotype-specific Serum Antibody Titers Measured by MOPA on Day 181
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by MOPA on Day 181 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Day 181 for the serotypes O1A, O2, O4, O6A, O15, O16, O18A, O25B and O75 was calculated as the ratio of titer values of serum antibody on Day 181 and pre-vaccination (on day 1) that is, Day 181/Day 1.
Time Frame: Baseline (Day 1, pre-vaccination) and Day 181
Reporting Status: Not Posted, anticipated posting 2025-12

41. Secondary Outcome: Cohort 2: Geometric Mean Ratio (GMR) of Serotype-specific Antibodies Measured by MOPA on Day 181
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by MOPA on Day 181 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O15, O16, O18A, O25B and O75 were determined in serum from collected blood samples by MOPA. GMR of fold change from baseline was calculated as the ratio of GMTs on Day 181 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination), Day 181
Reporting Status: Not Posted, anticipated posting 2025-12

42. Secondary Outcome: Cohort 2: Number of Participants With Serious Adverse Events (SAEs) Related to Study Vaccine or Study Procedure From Day 182 up to End of Study (Day 1826)
Description: as for outcome 28
Time Frame: From Day 182 up to end of study (Day 1826)
Reporting Status: Not Posted, anticipated posting 2025-12

43. Secondary Outcome: Cohort 2: Geometric Mean Titers (GMTs) of Serotype-specific Antibodies Against Specified Antigens Measured by Multiplex ECL Based Immunoassay on Day 366
Description: GMTs of serotype-specific antibodies as measured by ECL based immunoassay were reported. GMTs for the serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA were determined.
Time Frame: At Day 366
Reporting Status: Not Posted, anticipated posting 2025-12

44. Secondary Outcome: Cohort 2: Percentage of Participants With a >= 2-Fold and >=4-Fold Increase in Serotype-specific Serum Antibody Titers Measured by Multiplex ECL Based Immunoassay on Day 366
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by multiplex ECL based immunoassay on Day 366 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Day 366 for the serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA was calculated as the ratio of titer values of serum antibodies on Day 366 and pre-vaccination (on day 1) that is, Day 366/Day 1.
Time Frame: Baseline (Day 1, pre-vaccination) and Day 366
Reporting Status: Not Posted, anticipated posting 2025-12

45. Secondary Outcome: Cohort 2: Geometric Mean Ratio (GMR) of Serotype-specific Antibodies Measured by Multiplex ECL Based Immunoassay on Day 366
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by multiplex ECL based immunoassay on Day 366 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O8, O15, O16, O18A, O25B, O75 and EPA were determined in serum from collected blood samples by ECL based immunoassay. GMR of fold change from baseline was calculated as the ratio of GMTs on Day 366 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination), Day 366
Reporting Status: Not Posted, anticipated posting 2025-12

46. Secondary Outcome: Cohort 2: Geometric Mean Titers (GMTs) of Serotype-specific Antibodies Against Specified Antigens Measured by MOPA on Day 366
Description: as for outcome 39
Time Frame: At Day 366
Reporting Status: Not Posted, anticipated posting 2025-12

47. Secondary Outcome: Cohort 2: Percentage of Participants With a >= 2-Fold and >=4-Fold Increase in Serotype-specific Serum Antibody Titers Measured by MOPA on Day 366
Description: Percentage of participants with a >=2-fold and >=4-fold increase from baseline in serotype specific serum antibody titers as measured by MOPA on Day 366 was reported. The fold (>=2-fold and >=4-fold) increase from baseline to Day 366 for the serotypes O1A, O2, O4, O6A, O15, O16, O18A, O25B and O75 was calculated as the ratio of titer values of serum antibody on Day 366 and pre-vaccination (on day 1) that is, Day 366/Day 1.
Time Frame: Baseline (Day 1, pre-vaccination) and Day 366
Reporting Status: Not Posted, anticipated posting 2025-12

48. Secondary Outcome: Cohort 2: Geometric Mean Ratio (GMR) of Serotype-specific Antibodies Measured by MOPA on Day 366
Description: GMR of fold changes from baseline for serotype specific antibodies as measured by MOPA on Day 366 were reported. GMR for each antigen serotypes O1A, O2, O4, O6A, O15, O16, O18A, O25B and O75 were determined in serum from collected blood samples by MOPA. GMR of fold change from baseline was calculated as the ratio of GMTs on Day 366 and pre-vaccination (on Day 1).
Time Frame: Baseline (Day 1, pre-vaccination), Day 366
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: SAEs and All-Cause Mortality: Day 1 (post vaccination) up to Day 181; unsolicited AEs (not SAEs): Day 1 (post vaccination) up to 30 days; Solicited (local and systemic) AEs: up to 14 days post vaccination on Day 1 (from Day 1 up to Day 15)
Description: FAS included all participants with a study vaccine administration documented. Cohort 1 AEs were coded using MedDRA version 23.0 and Cohort 2 AEs were coded using MedDRA version 24.1.
Arm/Group | Cohort 1: Low Dose ExPEC10V | Cohort 1: Medium Dose ExPEC10V | Cohort 1: High Dose ExPEC10V | Cohort 1: ExPEC4V | Cohort 1: Prevnar 13 | Cohort 2: ExPEC10V High Dose | Cohort 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/102 | 0/104 | 0/52 | 0/54 | 0/278 | 0/138
Serious Adverse Events (participants affected / at risk) | 2/104 | 2/102 | 0/104 | 0/52 | 1/54 | 9/278 | 6/138
Other Adverse Events (participants affected / at risk) | 60/104 | 61/102 | 71/104 | 24/52 | 41/54 | 180/278 | 64/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Low Dose ExPEC10V (N=104) | Cohort 1: Medium Dose ExPEC10V (N=102) | Cohort 1: High Dose ExPEC10V (N=104) | Cohort 1: ExPEC4V (N=52) | Cohort 1: Prevnar 13 (N=54) | Cohort 2: ExPEC10V High Dose (N=278) | Cohort 2: Placebo (N=138)
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Enterococcal Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis Infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Low Dose ExPEC10V (N=104) | Cohort 1: Medium Dose ExPEC10V (N=102) | Cohort 1: High Dose ExPEC10V (N=104) | Cohort 1: ExPEC4V (N=52) | Cohort 1: Prevnar 13 (N=54) | Cohort 2: ExPEC10V High Dose (N=278) | Cohort 2: Placebo (N=138)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 4 | 1 | 0 | 3 | 3
Nausea (Gastrointestinal disorders) | 5 | 9 | 11 | 1 | 2 | 40 | 8
Erythema (General disorders) | 11 | 19 | 19 | 1 | 5 | 60 | 1
Fatigue (General disorders) | 21 | 29 | 24 | 8 | 13 | 98 | 31
Fever (General disorders) | 2 | 0 | 3 | 1 | 0 | 15 | 3
Injection Site Pruritus (General disorders) | 1 | 5 | 3 | 2 | 1 | 7 | 0
Pain/Tenderness (General disorders) | 46 | 52 | 60 | 15 | 39 | 132 | 20
Swelling (General disorders) | 9 | 15 | 14 | 2 | 2 | 44 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 4 | 1 | 3 | 3 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 7 | 10
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 0 | 0 | 7 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 36 | 37 | 10 | 21 | 84 | 23
Headache (Nervous system disorders) | 19 | 25 | 25 | 11 | 10 | 74 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03819049/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT03819049/SAP_001.pdf